CLINICAL TRIAL: NCT05713500
Title: Personality and Chronic Pain: a Comparative Study in Parkinson's Disease and Other Chronic Pain Conditions
Brief Title: Comparative Study of Personality in Parkinson's Disease Patients With Other Chronic Pain
Acronym: PSYCHO-PAIN
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0372
Record Dates: First submitted 2022-11-03; First posted 2023-02-06 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Chronic pain; personality
MeSH Terms: conditions — Parkinson Disease; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PD patients with chronic pain: Parkinsonian patient with pain
  Interventions: Other: TCI; Other: BPI; Other: CPAQ-8; Other: SF-MPQ; Other: King's Parkinson's Disease Pain Scale (KPPS); Other: Hospital Anxiety and Depression scale (HAD) questionary; Other: PCS; Other: ORT; Other: Social Support Questionnaire (SSQ6); Other: IPQ-R; Other: WCC-R
- PD patients without pain: Parkinsonian patient without pain
  Interventions: Other: TCI; Other: Hospital Anxiety and Depression scale (HAD) questionary; Other: ORT; Other: Social Support Questionnaire (SSQ6)
- non-PD patients with chronic pain: Non-PD with fibromyalgia and non-PD with chronic headache
  Interventions: Other: TCI; Other: BPI; Other: CPAQ-8; Other: SF-MPQ; Other: Hospital Anxiety and Depression scale (HAD) questionary; Other: PCS; Other: ORT

INTERVENTIONS:
Other: TCI — Temperament and character inventory
Other: BPI — Brief Pain Inventory
  Groups: PD patients with chronic pain; non-PD patients with chronic pain
Other: CPAQ-8 — Chronic Pain Acceptance Questionnaire-8
  Groups: PD patients with chronic pain; non-PD patients with chronic pain
Other: SF-MPQ — short-form McGill Pain Questionnaire
  Groups: PD patients with chronic pain; non-PD patients with chronic pain
Other: King's Parkinson's Disease Pain Scale (KPPS) — King's Parkinson's Disease Pain Scale
  Groups: PD patients with chronic pain
Other: Hospital Anxiety and Depression scale (HAD) questionary — Hospital Anxiety and Depression scale
Other: PCS — Pain Catastrophism Scale
  Groups: PD patients with chronic pain; non-PD patients with chronic pain
Other: ORT — Opioid Risk Tool
Other: Social Support Questionnaire (SSQ6) — Social Support Questionnaire (SSQ6) (score of availability and score of satisfaction)
  Groups: PD patients with chronic pain; PD patients without pain
Other: IPQ-R — Illness Perception Questionnaire Revised
  Groups: PD patients with chronic pain
Other: WCC-R — Ways of Coping Checklist Revised
  Groups: PD patients with chronic pain

SUMMARY:
The present study compare personality of Parkinson's Disease (PD) patients with chronic, PD patients without pain and non-parkinsonian patients with other chronic pain condition.

DETAILED DESCRIPTION:
The present study would like to compare personality dimensions from the Temperament and character inventory (TCI) in four groups of patients: PD patients with chronic pain related to PD, PD patients without pain and non-PD patients with chronic pain such as fibromyalgia or chronic headache. Our aim is to evaluate if PD patients with chronic pain related to PD have a different personality than PD patients without pain and to see if this personality is specific to PD.

ELIGIBILITY:
Inclusion Criteria:

* PD patients:

Patients having Parkinson's disease according to UNITED KINGDOM PARKINSON'S DISEASE SOCIETY BRAIN BANK (UKPDSBB) criteria

PD patients with chronic pain:

Patients with a pain VAS score ≥ 4 (mean VAS for the last week) Patients with a chronic pain since at least 3 months

PD patients without pain:

Patients with a pain VAS score < 3

* non PD patients:

Patients with chronic headache:

Patients with chronic headache according to the ICHD-3 beta criteria Patients with a chronic pain since at least 3 months

Patients with fibromyalgia:

Patients with fibromyalgia according to the criteria of the American College of Rheumatology 2016 (Wolfe et al., 2016) Patients with a pain VAS score ≥ 4 (mean VAS for the last week) Patients with a chronic pain since at least 3 months

* All patients:

Patient > 18 years old Patient able to give its free and informed consent Patient having a social security.

Exclusion Criteria:

* PD patients:

Patients presenting atypical Parkinson's syndrome Patients having a deep brain stimulation Patients presenting a cognitive decline evaluated by a Montreal Cognitive Assessment (MoCA) score inferior to 24

* All patients:

Patient having a psychiatric disease diagnosed according to the Diagnostic and Statistical Manual-V (DSM-V) criteria such as mood disorders, psychotic disorder… None ability to give its consent Patients unable to realize the tests provided in the context of this study Patients under supervision, curatorship, or legal guardian Patients non-affiliated to a social security Patients in exclusion period of another study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parkinsonian patients with and without chronic pain and non-parkinsonian patients with chronic pain such as fibromyalgia and headache
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
TCI personality dimensions between the two groups of patients | 24 months
  compare scores of the seven TCI personality dimensions between the two groups of parkinsonian patients with or without chronic pain related to PD. This will allow to determinate if PD patients with chronic pain related to PD have a different personality than PD patients without pain

SECONDARY OUTCOMES:
personality dimensions of the TCI and two-by-two analyses | 24 months
  compare personality dimensions of the TCI through two-by-two analyses between PD patients with chronic pain related to PD and patients presenting another chronic pain etiology:
  1) patients with fibromyalgia, 2) patients with chronic headache. This will allow to determinate if PD patients with chronic pain have a personality specific to their PD
association between personality the seven TCI and scores | 24 months
  determinate if there are some associations between the seven TCI personality dimensions of PD patients with chronic pain related to PD and different pain parameters:
  * the pain intensity evaluated with the Visual Analog Scale (VAS)
  * the functional discomfort evaluated with the Brief Pain Inventory (BPI)
  * the acceptation of pain evaluated with the Chronic Pain Acceptance questionnaire-8 (CPAQ-8)
  * the discriminative and affective components of pain evaluated with the Short-Form McGill Pain Questionnaire (SF-MPQ)
  * the level of catastrophism evaluated with the Pain Catastrophism Scale (PCS).
association between personality the seven TCI personality dimensions and different pain | 24 months
  determinate if there are some associations between the seven TCI personality dimensions of PD patients with chronic pain related to PD and different pain parameters:
  * the pain intensity evaluated with the VAS (Visual Analog Scale)
  * the functional discomfort evaluated with the BPI (Brief Pain Inventory)
  * the acceptation of pain evaluated with the CPAQ-8 (Chronic Pain Acceptance questionnaire-8)
  * the discriminative and affective components of pain evaluated with the SF-MPQ (short-form McGill Pain Questionnaire)
  * the level of catastrophism evaluated with the PCS (Pain Catastrophism Scale)
association of personality dimensions of the TCI and in other patients with chronic pain etiology | 24 months
  determinate if there are some associations between TCI personality dimensions and these same previous parameters (VAS, BPI, CPAQ-8, SF-MPQ, PCS and ORT) in other patients with chronic pain etiology: 1) first, in patients with fibromyalgia, 2) then, in patients with chronic headache
exploratory objective | 24 months
  determinate if there are some associations between TCI personality dimensions in PD patients with chronic pain related to PD and PD-specific pain evaluated by the King's Parkinson's Disease Pain Scale (KPPS)

CONTACTS AND LOCATIONS:
Overall Officials: Christine BREFEL-COURBON, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital (CHU de Toulouse), Toulouse, France

IPD SHARING:
Plan to Share IPD: No